CLINICAL TRIAL: NCT00051285
Title: ESSENTIAL Protocol No. My-021 and Protocol No. My-026, Each Titled: A Phase III, Randomized, Double-Blind, Multicenter, Parallel Group, Placebo-Controlled Study of Oral Enoximone vs. Placebo in Advanced Chronic Heart Failure Subjects
Brief Title: ESSENTIAL-"The Studies of Oral Enoximone Therapy in Advanced Heart Failure"
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESSENTIAL: My-021 and My-026
Record Dates: First submitted 2003-01-07; First posted 2003-01-09 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure, Congestive
Keywords: CHF; heart; failure; congestive; enoximone; phosphodiesterase; inhibitor
MeSH Terms: conditions — Heart Failure | interventions — Enoximone

ARMS (2):
- Enoximone (Experimental)
  Interventions: Drug: Enoximone
- Placebo (Placebo Comparator)
  Interventions: Drug: Enoximone placebo

INTERVENTIONS:
Drug: Enoximone — Participants receive oral enoximone
  Arms: Enoximone
Drug: Enoximone placebo — Participants receive placebo to match enoximone
  Arms: Placebo

SUMMARY:
To determine if low-dose enoximone therapy is an effective treatment for advanced chronic heart failure.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, multicenter, parallel group, placebo-controlled trial of oral enoximone in approximately 700 subjects with advanced chronic heart failure of either ischemic or nonischemic etiology receiving optimal conventional heart failure therapy.

Eligible subjects will be randomized in a 1:1 ratio to receive either enoximone or placebo at the Randomization Visit. The initial dose of study drug will be 25 mg t.i.d.(3xday) and will be administered immediately after randomization. Subjects who tolerate this initial dose will be continued on 25 mg t.i.d. for at least two weeks. After two weeks, eligible subjects will be titrated to 50 mg t.i.d. for the duration of the study.

ELIGIBILITY:
In order to be considered eligible subjects, the following entry criteria must be met:

* At least 18 years of age
* ischemic or nonischemic cardiomyopathy
* NYHA Class III or IV
* one hospitalization, or two outpatient visits, for the treatment of worsening heart failure within 12 months requiring the administration of I.V. heart failure therapy
* LVEDD >3.2 cm/m2 or >=6.0 cm
* LVEF of less than or equal to 30%
* concomitant treatment with optimal conventional heart failure therapy

Exclusion Criteria

Subjects who meet any one of the following criteria will be deemed ineligible for participation in the study:

Subjects on the following concomitant medications:

* Calcium antagonists other than amlodipine or felodipine
* Flecainide, encainide, propafenone, dofetilide or disopyramide
* Subjects receiving I.V. positive inotropic agents within seven days of the Screening Visit or Randomization Visit
* Subjects receiving a human B-type natriuretic peptide, including nesiritide, within seven days of the Screening Visit or Randomization Visit
* Subjects receiving oral or I.V. phosphodiesterase III inhibitors (PDEI III), including levosimendan and cilostazol, within seven days of the Screening Visit or Randomization Visit

  * Subjects with active hepatic (screening serum total bilirubin >= 3.0 mg/dl (>=51.3 umol/l), renal (screening serum creatinine >= 2.0 mg/dl (=178.8 umol/l)), hematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease
  * Subjects with a serum potassium <4.0 mEq/L or >5.5 mEq/L (<4.0 mmol/l or >5.5 mmol/l) at Randomization Visit
  * Subjects with a magnesium level of <1.0 mEq/L (<0.5 mmol/l) at Randomization Visit (Visit 0)
  * Subjects with a serum digoxin of >1.2 ng/ml (>1.5 nmol/l) or a serum digitoxin of >20 ng/ml (>26.2 nmol/l) at the Randomization Visit are excluded. A target serum digoxin level of <=1.0 ng/ml (<=1.3 nmol/l) is recommended

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800
Dates: Start 2002-02; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Time from randomization to all-cause mortality or cardiovascular hospitalization | Baseline to Month 6

SECONDARY OUTCOMES:
Change in Patient Global Assessment score | Baseline to Month 6
  Improvement in quality of life assessed by the Patient Global Assessment patient-reported outcomes tool
Change in Six-Minute Walk Test | Baseline to Month 6
  Improvement in quality of life assessed by the Six-Minute Walk Test, a measure of submaximal exercise tolerance